CLINICAL TRIAL: NCT05284994
Title: A Single-arm, Open-label, Multi-cohort, Multi-center Clinical Study on the Safety and Efficacy of TQ-B3525 Tablets Combined With Osimertinib in Subjects With Advanced Non-small Cell Lung Cancer
Brief Title: TQ-B3525 Tablets Combined With Osimertinib Mesylate Tablets in the Treatment of Advanced Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3525-Ib/II -01
Record Dates: First submitted 2022-03-03; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Nonsmall-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3525 Tablets + Osimertinib Mesylate Tablets. (Other): TQ-B3525 tablets combined with osimertinib mesylate tablets, 30 days as a treatment cycle.
  Interventions: Drug: TQ-B3525 Tablets, Osimertinib Mesylate Tablets

INTERVENTIONS:
Drug: TQ-B3525 Tablets, Osimertinib Mesylate Tablets — TQ-B3525 is a novel α/δ dual inhibitor PI3K kinase inhibitor. Osimertinib mesylate is a third-generation epidermal growth factor receptor inhibitor.

SUMMARY:
TQ-B3525 tablet is a new α/δ dual inhibitor phosphatidylinositol 3-kinase inhibitor developed by Chia Tai Tianqing pharmaceutical Group Co., Ltd. It can overcome the drug resistance problem caused by the up-regulation of phosphatidylinositol 3-kinase α subunit activity caused by the single inhibition of phosphatidylinositol 3-kinase δ subunit. This study is a single-arm, open-label, multi-cohort, multi-center clinical study of the safety and efficacy of TQ-B3525 tablets combined with osimertinib in subjects with advanced non-small cell lung cancer, aiming to evaluate TQ-B3525 tablets combined with osimertinib, the safety, tolerability, and efficacy of the treatment of patients with advanced non-small cell lung cancer who have failed epidermal growth factor receptor inhibitor therapy, while exploring the efficacy, resistance mechanism, and safety in the dose escalation phase biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* 1 Aged 18 to 75 years old, and gender is not limited.
* 2 The eastern cooperative oncology group（ECOG）score is 0 to 1, and the expected survival time is greater than or equal to 12 weeks.
* 3 Subjects with histologically or cytologically confirmed non-small cell lung cancer (NSCLC) and stage IIIB-IV (according to the 8th edition of the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer Classification).
* 4 The enrollment requirements for the dose escalation phase are as follows:

  1. Patients who have failed previous standard therapy, including disease progression or toxicity intolerance, or who are clinically unsuitable or unacceptable, or who refuse to receive standard therapy.
  2. The test report can reflect the presence of epidermal growth factor receptor (EGFR) sensitive mutations when the subjects were enrolled in this trial.
  3. Requirements for meeting the epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) treatment failure criteria:

     1. Subjects without T790M mutation after receiving first- or second-generation epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) treatment resistance in the past; or subjects who have previously received third-generation epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) treatment resistance.
     2. According to the definition of response evaluation criteria in solid tumors Recist version 1.1 (Recist 1.1) criteria, disease progression occurs after continuous epidermal growth factor receptor- -tyrosine kinase inhibitor treatment for at least 1 month.
     3. No other systemic therapy between discontinuation of epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) and initiation of new therapy.
* 5 The enrollment requirements for Cohort 1 in the dose expansion phase are as follows:

  1. failure of previous standard therapy, including disease progression or toxicity intolerance, or clinical inappropriateness/inability to accept/refusal to receive standard therapy.
  2. There is a sensitive epidermal growth factor receptor（EGFR） mutation, and previous reports have confirmed that it is accompanied by a gene abnormality in the PI3K signaling pathway.
  3. Requirements for meeting the epidermal growth factor receptor-tyrosine kinase inhibitor（EGFR-TKI）treatment failure criteria:

     1. Subjects without T790M mutation after receiving first- or second-generation epidermal growth factor receptor-tyrosine kinase inhibitor（EGFR-TKI） treatment resistance in the past; or subjects who have previously received third-generation epidermal growth factor receptor-tyrosine kinase inhibitor（EGFR-TKI）treatment resistance.
     2. According to the definition of response evaluation criteria in solid tumors Recist version 1.1(Recist 1.1)criteria, disease progression occurs after continuous epidermal growth factor receptor-tyrosine kinase inhibitor(EGFR-TKI) treatment for at least 1 month.
     3. No other systemic therapy between discontinuation of epidermal growth factor receptor-tyrosine kinase inhibitor（EGFR-TKI）and initiation of new therapy.
* 6 Enrollment requirements for Cohort 2 in the dose expansion phase are as follows:

  1. failure of previous standard therapy, including disease progression or toxicity intolerance, or clinically inappropriate, or unacceptable, or refusal to receive standard therapy.
  2. There is a sensitive epidermal growth factor receptor（EGFR） mutation, and previous reports have confirmed that there is no abnormality in the PI3K signaling pathway, and the report can reflect the gene status of the subjects when they are enrolled in this trial.
  3. Meet the following definitions for epidermal growth factor receptor-tyrosine kinase inhibitor（EGFR-TKI）treatment failure:

     1. Subjects without T790M mutation after receiving first- or second-generation epidermal growth factor receptor-tyrosine kinase inhibitor（EGFR-TKI） treatment resistance in the past; or subjects who have previously received third-generation epidermal growth factor receptor-tyrosine kinase inhibitor（EGFR-TKI）treatment resistance.
     2. According to the definition of response evaluation criteria in solid tumors Recist version 1.1（Recist 1.1）criteria, disease progression occurs after continuous epidermal growth factor receptor-tyrosine kinase inhibitor（EGFR-TKI） treatment for at least 1 month.
     3. No other systemic therapy between discontinuation of epidermal growth factor receptor-tyrosine kinase inhibitor（EGFR-TKI）and initiation of new therapy.
* 7 The enrollment requirements for Cohort 3 in the dose expansion phase are as follows.

  1. Have not received any systemic therapy for locally advanced or metastatic NSCLC before.
  2. There are epidermal growth factor receptor（EGFR） sensitive mutations, and the test report can reflect the gene status of the subjects when they are enrolled in this trial.
* 8 At the time of screening, according to response evaluation criteria in solid tumors Recist version 1.1（Recist 1.1）criteria, the patient has at least one measurable target lesion.
* 9 Inspections during the screening period shall meet the following conditions:

  1. The absolute value of neutrophils (ANC) is greater than or equal to 1.5×109/L.
  2. Platelet count (PLT) greater than or equal to 75×109/L.
  3. Hemoglobin is greater than or equal to 90g/L.
  4. The total blood bilirubin is less than or equal to 1.5 times the upper limit of normal（ULN）. If it is a subject with Gilbert syndrome, the total blood bilirubin is less than or equal to 3×upper limit of normal（ULN）.
  5. Serum creatinine (Cr) is less than or equal to 1.5×upper limit of normal（ULN）, or creatinine clearance rate is greater than or equal to 60ml/min.
  6. alanine aminotransferase（ALT）and aspartate aminotransferase（AST）are less than or equal to 2.5 times upper limit of normal（ULN）. If there is liver metastasis, alanine aminotransferase（ALT）and aspartate aminotransferase（AST）can be relaxed to the corresponding 5 times upper limit of normal（ULN）.
  7. Coagulation function tests must meet the following criteria: prothrombin time (PT), activated partial thromboplastin time (APTT), and international normalized ratio (INR) are all less than or equal to 1.5 times the upper limit of normal (ULN) coagulation therapy) .
  8. Doppler ultrasound: left ventricular ejection fraction (LVEF) greater than or equal to 50%.
* 10 The subjects voluntarily participated in this study and signed the informed consent.

Exclusion Criteria:

* 1 There are contraindications to Osimertinib Mesylate Tablets administration.
* 2 Other malignant tumors that have occurred or are currently at the same time within 3 years, except for cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumor.
* 3 The subject has received PI3K inhibitor treatment in the past.
* 4 Subjects who have received other systemic anti-tumor drugs within 3 weeks before the first dose, or who are still within the in 5 half-life period of the drug.
* 5 Received any major surgical treatment within 4 weeks before the first dosage.
* 6 Received any previous radiotherapy for curative purposes within 2 weeks before the first drug.
* 7 Unrelieved toxic reactions higher than common terminology criteria for adverse events （CTC AE）grade 1 due to any previous treatment, excluding alopecia.
* 8 The subjects had active serious viral, or bacterial, or fungal infections within 4 weeks before the first administration.
* 9 One of the following conditions of grade II or above occurred within 6 months before the first medication: myocardial infarction, severe or unstable angina pectoris, coronary or peripheral artery bypass grafting, cerebrovascular accident, including transient cerebral ischemia attack, as well as deep vein thrombosis or pulmonary embolism.
* 10 Current uncontrolled congestive heart failure.
* 11 Currently there is persistent arrhythmia greater than or equal to grade II, any degree of uncontrolled atrial fibrillation or QTc interval greater than 480 ms.
* 12 Subjects with unsatisfactory blood pressure control, that is, subjects with systolic blood pressure greater than or equal to 150 mmHg and diastolic blood pressure greater than or equal to 100 mmHg.
* 13 Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage.
* 14 Type I and type II diabetes, in addition to only taking exercise and diet control, or only needing a single oral hypoglycemic drug to stably control blood sugar, and fasting blood sugar less than 7.0 mmol/L and glycosylated hemoglobin (HbA1c) less than 7.0 during the screening period % of subjects with type II diabetes.
* 15 Presence of interstitial lung disease, severely impaired lung function, severe pulmonary fibrosis, radiation pneumonitis, history of drug-induced lung disease, and evidence of active pulmonary inflammation on chest computed tomography (CT) findings during screening.
* 16 Subjects with a history of immunodeficiency, including but not limited to HIV-positive or other acquired, congenital immunodeficiency diseases, or subjects with active autoimmune diseases or a history of autoimmune diseases.
* 17 There is currently a severe and unstable central nervous system metastasis. Note: Patients with no or mildly symptomatic central nervous system（CNS）metastases can be included. Whole brain radiation or gamma knife therapy received due to central nervous system（CNS）metastases must be completed 14 days before the first dose and clinically stable.
* 18 When virological testing during the screening period shows any of the following:

  1. hepatitis B surface antigen（HBsAg）positive and hepatitis B virus Deoxyribonucleic acid（HBV-DNA）exceeding the upper limit of normal or hepatitis B virus Deoxyribonucleic acid（HBV-DNA）exceeding 1000copies/ml.
  2. Anti- hepatitis C virus（HCV）positive and hepatitis C virus（HCV）ribonucleic acid（RNA）positive or beyond the upper limit of normal.
* 19 People with multiple factors that affect oral administration and drug absorption, such as inability to swallow, post gastrointestinal resection, ulcerative colitis, symptomatic or inflammatory bowel disease, chronic diarrhea and intestinal obstruction and other gastrointestinal diseases.
* 20 Women of childbearing age have a positive pregnancy test before administration of the study drug, or who cannot guarantee to take effective contraceptive measures during the study period, and men cannot guarantee to take effective contraceptive measures during the study period.
* 21 Any other circumstances that are judged by the investigator to be incapable of being included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Baseline time to increase chemotherapy drug dose to toxicity intolerance, up to 5 weeks.
  Some major toxic and side effects of drugs are the main reasons for restricting the continued increase in the dose of chemotherapeutic drugs. These toxic and side effects are the dose-limiting toxicity of chemotherapeutic drugs.
Objective response rate (ORR) | From date of first medication until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  Objective response rate refers to the proportion of patients whose tumor shrinkage reaches a certain amount and maintains it for a certain period of time, including complete response (CR)+ partial response (PR) cases.

SECONDARY OUTCOMES:
Progression-Free-Survival (PFS) | From date of first medication until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  Progression-free survival refers to the time span from the start of tumor treatment to the occurrence of secondary growth of the tumor. It means that the tumor basically does not progress at this stage.
Disease Control Rate (DCR) | From date of first medication until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  Disease control rate refers to the percentage of cases with remission and stable disease after treatment in the total number of evaluable cases.
Overall Survival (OS) | From date of first medication until the date of death from any cause，an average of 5 years.
  Overall survival is the time from first medication to death from any cause.
Duration of disease remission | Tumors were first assessed as complete response (CR) or partial response (PR) from the date of disease progression or death, whichever occurred first. Through study completion, an average of 1 year.
  Duration of disease response refers to the time from the first tumor assessment as complete response (CR) or partial response (PR) to the first assessment as PD or death from any cause.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Sun-Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Southern Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - The Second People's Hospital of Guangdong Province, Guanzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Affiliated Hospital Of Guangdong Medical University, Zhanjiang, Guangdong